CLINICAL TRIAL: NCT06487325
Title: Clinical Study of Ultrasound-derived Fat Fraction to Assess Metabolic Dysfunction-Associated Steatotic Liver Disease in Obese Population
Brief Title: A Clinical Study of Ultrasound-derived Fat Fraction to Assess Metabolic Dysfunction-Associated Steatotic Liver Disease
Status: Completed | Type: Observational
Sponsor: Ma Zhe (Other)
Responsible Party: Sponsor-Investigator, Ma Zhe, Director of Ultrasound, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2024(014)
Record Dates: First submitted 2024-06-26; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group S1: Liver biopsy showed mild fatty liver
- Group S2: Liver biopsy showed moderate fatty liver
- Group S3: Liver biopsy showed severe fatty liver

SUMMARY:
Aims: To evaluate the diagnostic performance of ultrasound-derived fat fraction (UDFF) in assessing the degree of hepatic steatosis in an obese population, with liver biopsy as reference standard.

Materials and methods: Obese individuals, who were found to have fatty liver by B-mode ultrasound and underwent UDFF measurement, along with liver biopsy results, were retrospectively selected from The First Affiliated Hospital of Shandong First Medical University.The inclusion criteria were as follows: (1) BMI over 30 kg/m²; (2) diffuse fatty liver or inhomogeneous fatty liver diagnosed by conventional B-mode ultrasound; (3) serologic test results were available. The exclusion criteria include: (1) patients who have undergone liver resection or have liver space-occupying lesions; (2) pregnant women; (3) patients with incomplete medical history data.

ELIGIBILITY:
Inclusion Criteria:

* BMI over 30 kg/m²
* diffuse fatty liver or inhomogeneous fatty liver diagnosed by conventional B-mode ultrasound
* serologic test results were available

Exclusion Criteria:

* patients who have undergone liver resection or have liver space-occupying lesions
* pregnant women
* patients with incomplete medical history data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese individuals, who were found to have fatty liver by B-mode ultrasound and underwent UDFF measurement, along with liver biopsy results, were retrospectively selected from The First Affiliated Hospital of Shandong First Medical University
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-04-29 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
UDFF values | up to 1 year
  During the examination, the DAX probe was positioned in the right intercostal space, and the UDFF mode was selected to place a fixed-size region of interest (ROI) vertically in the right lobe of the liver, 1.5 cm away from the liver capsule, avoiding the intrahepatic duct structure. Measurements were acquired after the patient maintained a calm breathing pattern, and the system automatically determined the shear wave velocity (Vs), elastic modulus (E), and UDFF values.

SECONDARY OUTCOMES:
SWE values | up to 1 year
  The auto-SWE values were collected simultaneously when using UDFF mode, and the SWE and pSWE values were collected 10 times with 5C1 and DAX probes, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- QianfoshanH, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Lack of resources or infrastructure: Sharing IPDs requires resources and infrastructure to ensure data security, manage access requests and provide necessary documentation. Currently these resources are not well developed, so it may be difficult to share IPDs.